CLINICAL TRIAL: NCT00117832
Title: Nasal Ocular Reflexes Contribute to Eye Symptoms in Patients With Allergic Rhinitis
Brief Title: Nasal Ocular Reflexes Contribute to Eye Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 13716A
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Azelastine nasal spray

SUMMARY:
Eye symptoms of tearing, redness and itching frequently occur in patients with allergic rhinitis or hayfever. The purpose of this trial is to study whether placing an allergen (a substance that causes allergies) directly in your nose can cause you to have eye symptoms as well as nasal symptoms.

DETAILED DESCRIPTION:
Symptoms of conjunctivitis (tearing, redness and itching) frequently occur in patients with allergic rhinitis. The pathophysiology underlying these symptoms remains to be elucidated. The symptoms probably arise via a combination of mechanisms including direct contact of natural pollen with the conjunctiva and reflex mechanisms originating in the nose.

Pollen exposure can result from direct hand transfer of pollen to the conjunctiva or, conceivably, from the forceful blowing of air, containing nasal secretions with antigen, up the nasolacrimal duct. The latter mechanism would be considered extremely unlikely because of the location of the nasolacrimal duct under the inferior turbinate (the duct's location is in an area with little pollen exposure) and the considerable force of air needed to cause reverse flow in the duct. The latter would also be true for topically applied intranasal drugs reaching the conjunctiva via the nasolacrimal duct, whereas the administration of medications to the conjunctiva frequently results in these medications reaching the nose via the nasolacrimal duct.

In support of direct contact of pollen as a source of ocular symptoms in patients with allergic rhinitis is the observation that pollen can be washed out of the conjunctiva on windy days, although the amount is 10 fold less than the amount of pollen recovered simultaneously from the nose. Additionally, beginning with Noon in the early 1900s, and subsequently shown by others, direct conjunctival challenges induce ocular symptoms. Thus, direct contact is a plausible explanation, but its relative contribution to eye symptoms in allergic rhinitis is unknown. Since topical intranasal steroids are known to reduce eye symptoms and the chance of them reaching the eye by systemic absorption or directly when administered intranasally are very slim, the investigators would postulate that direct allergen contact at the conjunctiva is a small contributor to the overall ocular symptom complex.

Reflex mechanisms within the nose have been shown to occur universally in response to nasal challenge with antigen. Nasal challenge with antigen induces a reflex in the contralateral nasal cavity, known as the nasonasal reflex. This reflex can also be initiated by nasal challenge with cold, dry air and histamine. The contralateral response to antigen, cold dry air and histamine is blocked by topical anticholinergic agents applied to the contralateral side, suggesting that the efferent limb is parasympathetically mediated. Histamine is only released on the side of challenge with antigen but oral H1 antihistamines reduce the contralateral response to unilateral nasal allergen challenge, suggesting that histamine contributes to the initiation of the reflex. The eye is richly innervated by parasympathetic nerves which enter the eye after running in conjunction with the parasympathetic input to the nasal cavity. The investigators, therefore, hypothesize that the conjunctiva will respond to nasal allergen in a manner similar to the contralateral nasal cavity.

Purpose: The investigators will study whether antigen-induced nasal reflexes cause eye symptoms. The investigators suspect that reflexes occur between the nose and the eye, and contribute substantially to eye symptoms in allergic patients during the allergy season. The investigators propose to demonstrate that nasal challenge with antigen leads to increased lacrimation.

ELIGIBILITY:
Inclusion Criteria:

* History of grass and/or ragweed allergic rhinitis.
* Positive skin test to grass and/or ragweed antigen.
* Positive response to screening nasal challenge.

Exclusion Criteria:

* Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
* Pregnant or lactating women.
* Upper respiratory infection within 14 days of study start.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Amount of eye secretions collected on Schirmer strips following antigen challenge

SECONDARY OUTCOMES:
Amount of eye secretions collected on Schirmer strips following antigen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Philip G, Nayak AS, Berger WE, Leynadier F, Vrijens F, Dass SB, Reiss TF. The effect of montelukast on rhinitis symptoms in patients with asthma and seasonal allergic rhinitis. Curr Med Res Opin. 2004 Oct;20(10):1549-58. doi: 10.1185/030079904x3348. PMID 15462688
- [Background] Yanez A, Rodrigo GJ. Intranasal corticosteroids versus topical H1 receptor antagonists for the treatment of allergic rhinitis: a systematic review with meta-analysis. Ann Allergy Asthma Immunol. 2002 Nov;89(5):479-84. doi: 10.1016/S1081-1206(10)62085-6. PMID 12452206
- [Background] Gray RD, Haggart K, Lee DK, Cull S, Lipworth BJ. Effects of butterbur treatment in intermittent allergic rhinitis: a placebo-controlled evaluation. Ann Allergy Asthma Immunol. 2004 Jul;93(1):56-60. doi: 10.1016/S1081-1206(10)61447-0. PMID 15281472
- [Background] Hampel F Jr, Howland W 3rd, Van Bavel J, Ratner P. A randomized, double-blind, placebo-controlled study comparing the efficacy and safety of ebastine (20 mg and 10 mg) to loratadine 10 mg once daily in the treatment of seasonal allergic rhinitis. J Investig Allergol Clin Immunol. 2004;14(1):56-63. PMID 15160443
- [Background] Shahar E, Hassoun G, Pollack S. Effect of vitamin E supplementation on the regular treatment of seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2004 Jun;92(6):654-8. doi: 10.1016/S1081-1206(10)61432-9. PMID 15237767
- [Background] van Adelsberg J, Philip G, Pedinoff AJ, Meltzer EO, Ratner PH, Menten J, Reiss TF; Montelukast Fall Rhinitis Study Group. Montelukast improves symptoms of seasonal allergic rhinitis over a 4-week treatment period. Allergy. 2003 Dec;58(12):1268-76. doi: 10.1046/j.1398-9995.2003.00261.x. PMID 14616102
- [Background] Remberg P, Bjork L, Hedner T, Sterner O. Characteristics, clinical effect profile and tolerability of a nasal spray preparation of Artemisia abrotanum L. for allergic rhinitis. Phytomedicine. 2004 Jan;11(1):36-42. doi: 10.1078/0944-7113-00350. PMID 14971719
- [Background] Kirchhoff CH, Kremer B, Haaf-von Below S, Kyrein HJ, Mosges R. Effects of dimethindene maleate nasal spray on the quality of life in seasonal allergic rhinitis. Rhinology. 2003 Sep;41(3):159-66. PMID 14579656
- [Background] Lumry W, Hampel F, LaForce C, Kiechel F, el-Akkad T, Murray JJ. A comparison of once-daily triamcinolone acetonide aqueous and twice-daily beclomethasone dipropionate aqueous nasal sprays in the treatment of seasonal allergic rhinitis. Allergy Asthma Proc. 2003 May-Jun;24(3):203-10. PMID 12866325
- [Background] van Adelsberg J, Philip G, LaForce CF, Weinstein SF, Menten J, Malice MP, Reiss TF; Montelukast Spring Rhinitis Investigator Group. Randomized controlled trial evaluating the clinical benefit of montelukast for treating spring seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2003 Feb;90(2):214-22. doi: 10.1016/S1081-1206(10)62144-8. PMID 12602669
- [Background] Nayak AS, Philip G, Lu S, Malice MP, Reiss TF; Montelukast Fall Rhinitis Investigator Group. Efficacy and tolerability of montelukast alone or in combination with loratadine in seasonal allergic rhinitis: a multicenter, randomized, double-blind, placebo-controlled trial performed in the fall. Ann Allergy Asthma Immunol. 2002 Jun;88(6):592-600. doi: 10.1016/S1081-1206(10)61891-1. PMID 12086367
- [Background] Wilson AM, Orr LC, Coutie WJ, Sims EJ, Lipworth BJ. A comparison of once daily fexofenadine versus the combination of montelukast plus loratadine on domiciliary nasal peak flow and symptoms in seasonal allergic rhinitis. Clin Exp Allergy. 2002 Jan;32(1):126-32. doi: 10.1046/j.0022-0477.2001.01252.x. PMID 12002729
- [Background] Kilpelainen M, Terho EO, Helenius H, Koskenvuo M. Validation of a new questionnaire on asthma, allergic rhinitis, and conjunctivitis in young adults. Allergy. 2001 May;56(5):377-84. doi: 10.1034/j.1398-9995.2001.056005377.x. PMID 11350300
- [Background] Ratner PH, Lim JC, Georges GC. Comparison of once-daily ebastine 20 mg, ebastine 10 mg, loratadine 10 mg, and placebo in the treatment of seasonal allergic rhinitis. The Ebastine Study Group. J Allergy Clin Immunol. 2000 Jun;105(6 Pt 1):1101-7. doi: 10.1067/mai.2000.105525. PMID 10856142
- [Background] Van Cauwenberge P, Juniper EF. Comparison of the efficacy, safety and quality of life provided by fexofenadine hydrochloride 120 mg, loratadine 10 mg and placebo administered once daily for the treatment of seasonal allergic rhinitis. Clin Exp Allergy. 2000 Jun;30(6):891-9. doi: 10.1046/j.1365-2222.2000.00914.x. PMID 10848909
- [Background] Meltzer EO, Malmstrom K, Lu S, Prenner BM, Wei LX, Weinstein SF, Wolfe JD, Reiss TF. Concomitant montelukast and loratadine as treatment for seasonal allergic rhinitis: a randomized, placebo-controlled clinical trial. J Allergy Clin Immunol. 2000 May;105(5):917-22. doi: 10.1067/mai.2000.106040. PMID 10808172
- [Background] Hadley JA. Evaluation and management of allergic rhinitis. Med Clin North Am. 1999 Jan;83(1):13-25. doi: 10.1016/s0025-7125(05)70084-5. PMID 9927957
- [Background] Yang WH, Dolovich J, Drouin MA, Keith P, Haddon J, Jennings B. Comparison of budesonide Turbuhaler with budesonide aqua in the treatment of seasonal allergic rhinitis. Rhinocort Study Group. Can Respir J. 1998 Nov-Dec;5(6):455-60. doi: 10.1155/1998/639710. PMID 10070173
- [Background] Stern MA, Dahl R, Nielsen LP, Pedersen B, Schrewelius C. A comparison of aqueous suspensions of budesonide nasal spray (128 micrograms and 256 micrograms once daily) and fluticasone propionate nasal spray (200 micrograms once daily) in the treatment of adult patients with seasonal allergic rhinitis. Am J Rhinol. 1997 Jul-Aug;11(4):323-30. doi: 10.2500/105065897781446658. PMID 9292184
- [Background] Simola M, Boss I, Holopainen E, Malmberg H, Ruoppi P, Seppa J, Siivonen L, Suonpaa J, Piepponen T. Astemizole in combination with pseudoephedrine in the treatment of seasonal allergic rhinitis. Rhinology. 1996 Mar;34(1):21-3. PMID 8739863
- [Background] Pedersen B, Dahl R, Richards DH, Jacques LA, Larsen BB, Pichler W, Nykanen KN. Once daily fluticasone propionate aqueous nasal spray controls symptoms of most patients with seasonal allergic rhinitis. Allergy. 1995 Oct;50(10):794-9. doi: 10.1111/j.1398-9995.1995.tb05051.x. PMID 8607560
- [Background] Settipane G, Korenblat PE, Winder J, Lumry W, Murphree J, Alderfer VB, Simpson B, Smith JA. Triamcinolone acetonide Aqueous nasal spray in patients with seasonal ragweed allergic rhinitis: a placebo-controlled, double-blind study. Clin Ther. 1995 Mar-Apr;17(2):252-63. doi: 10.1016/0149-2918(95)80023-9. PMID 7614525
- [Background] Darnell R, Pecoud A, Richards DH. A double-blind comparison of fluticasone propionate aqueous nasal spray, terfenadine tablets and placebo in the treatment of patients with seasonal allergic rhinitis to grass pollen. Clin Exp Allergy. 1994 Dec;24(12):1144-50. doi: 10.1111/j.1365-2222.1994.tb03320.x. PMID 7889428
- [Background] Loth S, Bende M. Effect of nasal anaesthesia on lacrimal function after nasal allergen challenge. Clin Exp Allergy. 1994 Apr;24(4):375-6. doi: 10.1111/j.1365-2222.1994.tb00249.x. PMID 8039024
- [Background] Dolovich J, O'Connor M, Stepner N, Smith A, Sharma RK. Double-blind comparison of intranasal fluticasone propionate, 200 micrograms, once daily with 200 micrograms twice daily in the treatment of patients with severe seasonal allergic rhinitis to ragweed. Ann Allergy. 1994 May;72(5):435-40. PMID 8179230
- [Background] Bousquet J, Chanal I, Alquie MC, Charpin D, Didier A, Germouty J, Greillier P, Ickovic MH, Maria Y, Montane F, et al. Prevention of pollen rhinitis symptoms: comparison of fluticasone propionate aqueous nasal spray and disodium cromoglycate aqueous nasal spray. A multicenter, double-blind, double-dummy, parallel-group study. Allergy. 1993 Jul;48(5):327-33. doi: 10.1111/j.1398-9995.1993.tb02401.x. PMID 8368459
- [Background] Frolund L. Efficacy of an oral antihistamine, loratadine, as compared with a nasal steroid spray, beclomethasone dipropionate, in seasonal allergic rhinitis. Clin Otolaryngol Allied Sci. 1991 Dec;16(6):527-31. doi: 10.1111/j.1365-2273.1991.tb00965.x. PMID 1685945
- [Background] Juniper EF, Guyatt GH, O'Byrne PM, Viveiros M. Aqueous beclomethasone diproprionate nasal spray: regular versus "as required" use in the treatment of seasonal allergic rhinitis. J Allergy Clin Immunol. 1990 Sep;86(3 Pt 1):380-6. doi: 10.1016/s0091-6749(05)80101-0. PMID 2212409
- [Background] Frolund L, Etholm B, Irander K, Johannessen TA, Odkvist L, Ohlander B, Weeke B. A multicentre study of loratadine, clemastine and placebo in patients with perennial allergic rhinitis. Allergy. 1990 May;45(4):254-61. doi: 10.1111/j.1398-9995.1990.tb00493.x. PMID 2143361
- [Background] Johansen LV, Bjerrum P, Illum P. Treatment of seasonal allergic rhinitis--a double blind, group comparative study of terfenadine and dexchlorpheniramine. Rhinology. 1987 Mar;25(1):35-40. PMID 2883715
- [Background] Borum P, Gronborg H, Mygind N. Seasonal allergic rhinitis and depot injection of a corticosteroid. Evaluation of the efficacy of medication early and late in the season based on detailed symptom recording. Allergy. 1987 Jan;42(1):26-32. doi: 10.1111/j.1398-9995.1987.tb02183.x. PMID 3551670
- [Background] Wood SF. Oral antihistamine or nasal steroid in hay fever: a double-blind double-dummy comparative study of once daily oral astemizole vs twice daily nasal beclomethasone dipropionate. Clin Allergy. 1986 May;16(3):195-201. doi: 10.1111/j.1365-2222.1986.tb00766.x. PMID 3087656
- [Background] Orgel HA, Meltzer EO, Kemp JP, Welch MJ. Clinical, rhinomanometric, and cytologic evaluation of seasonal allergic rhinitis treated with beclomethasone dipropionate as aqueous nasal spray or pressurized aerosol. J Allergy Clin Immunol. 1986 Jun;77(6):858-64. doi: 10.1016/0091-6749(86)90384-2. PMID 3711553
- [Background] Backhouse CI, Finnamore VP, Gosden CW. Treatment of seasonal allergic rhinitis with flunisolide and terfenadine. J Int Med Res. 1986;14(1):35-41. PMID 3082694
- [Background] Beswick KB, Kenyon GS, Cherry JR. A comparative study of beclomethasone dipropionate aqueous nasal spray with terfenadine tablets in seasonal allergic rhinitis. Curr Med Res Opin. 1985;9(8):560-7. doi: 10.1185/03007998509109635. PMID 2863090
- [Background] Schaaf L, Hendeles L, Weinberger M. Suppression of seasonal allergic rhinitis symptoms with daily hydroxyzine. J Allergy Clin Immunol. 1979 Feb;63(2):129-33. doi: 10.1016/0091-6749(79)90203-3. PMID 365920
- [Background] Cockcroft DW, MacCormack DW, Newhouse MT, Hargreave FE. Beclomethasone dipropionate aerosol in allergic rhinitis. Can Med Assoc J. 1976 Sep 18;115(6):523-6. PMID 782679
- [Background] Lofkvist T, Svensson G. An open assessment of becotide (beclomethasone dipropionate) nasal spray in seasonal allergic rhinitis. Acta Allergol. 1975 Oct;30(4):227-38. doi: 10.1111/j.1398-9995.1975.tb01345.x. PMID 1106108
- [Derived] Baroody FM, Foster KA, Markaryan A, deTineo M, Naclerio RM. Nasal ocular reflexes and eye symptoms in patients with allergic rhinitis. Ann Allergy Asthma Immunol. 2008 Mar;100(3):194-9. doi: 10.1016/S1081-1206(10)60442-5. PMID 18426137